CLINICAL TRIAL: NCT01339689
Title: A Proof-of-Concept, Double-blind, Randomized, Placebo-controlled Study of Ganaxolone in Posttraumatic Stress Disorder
Brief Title: Ganaxolone in Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Collaborators: INTRuST, Post-Traumatic Stress Disorder - Traumatic Brain Injury Clinical Consortium (Other); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-0700
Record Dates: First submitted 2011-04-19; First posted 2011-04-21 (Estimated); Results first posted 2022-12-29 (Actual); Last update posted 2022-12-29 (Actual); Status verified 2022-11

CONDITIONS: PTSD
Keywords: PTSD; Posttraumatic Stress Disorder; pharmacotherapy; ganaxolone
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — ganaxolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ganaxolone (Experimental): active
  Interventions: Drug: Ganaxolone
- Placebo (Placebo Comparator): non-active
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ganaxolone — 200-600 mg bid, capsules, up to 12 weeks
  Other Names: GNX
  Arms: Ganaxolone
Drug: Placebo — capsules, bid, up to 12 weeks
  Other Names: PBO
  Arms: Placebo

SUMMARY:
This Phase 2 proof-of-concept study is a double-blind, randomized, placebo-controlled, 15-week investigation of ganaxolone versus placebo for the treatment of Posttraumatic Stress Disorder (PTSD). Up to 120 participants will be enrolled and randomized to receive either ganaxolone or placebo for 6 weeks. After 6 weeks of randomized treatment all participants will continue for 6 weeks on ganaxolone. The aim of the study is to assess the efficacy of ganaxolone compared to placebo for the treatment of PTSD symptoms after 6 weeks of treatment using the Clinician-Administered PTSD Rating Scale (CAPS). The second aim of the study is to evaluate the safety and tolerability of ganaxolone in the PTSD population.

ELIGIBILITY:
Key Inclusion Criteria:

* Veteran or civilian adult outpatients 18-55 years of age, with primary PTSD as defined by Diagnostic and Statistical manual of Mental Disorders-IV (DSM-IV) for at least 6 months
* Must be in general good health-confirmed by medical history, physical examination, and screening laboratory results
* Negative urine drug screen for drugs of abuse
* Negative urine pregnancy test for females of childbearing potential
* Sexually active participants are required to use a medically acceptable form of birth control

Key Exclusion Criteria

* Clinically unstable medical disease; progressive CNS disorder/disease; history of seizures (except childhood febrile seizure); moderate or severe traumatic brain injury (TBI)
* Females who are pregnant or currently breast feeding
* Current or past psychotic disorder, bipolar Type I disorder, or dementia
* Participants with recent drug abuse or dependency (excluding nicotine and caffeine)
* Participants unwilling to comply with the required alcohol prohibition during the trial
* Current suicidal or homicidal ideation necessitating intervention, and those with a history of suicide attempt in the past 10 years
* Participants with pending litigation related to the traumatic event
* Participants who are unwilling to withhold grapefruit or grapefruit juice for the duration of the study
* Participants receiving psychotherapy without a stable paradigm for at least 3 months
* Non-English speaking participants.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Marx, MD, MA, Principal Investigator — Duke University Medical Center and Durham VA Medical Center; Ann Rasmusson, MD, Principal Investigator — Boston University School of Medicine Research Affiliate, National Center for PTSD
Locations (8):
- United States (8):
  - VA San Diego Healthcare System/ University of California, San Diego, San Diego, California
  - Washington DC VA Medical Center/ Uniformed Services University of the Health Services, Washington D.C., District of Columbia
  - VA Boston Healthcare Services/ Spaulding Rehabilitation Hospital, Boston, Massachusetts
  - Manchester VA Medical Center/ Dartmouth College, Manchester, New Hampshire
  - Durham VA Medical Center /Duke University Medical Center, Durham, North Carolina
  - Cincinnati VA Medical Center/ University of Cincinnati, Cincinnati, Ohio
  - Charleston VA Medica Center/ Medical University of South Carolina, Charleston, South Carolina
  - White River Junction VA Medical Center/ Dartmouth College, White River Junction, Vermont

REFERENCES:
- [Derived] Rasmusson AM, Marx CE, Jain S, Farfel GM, Tsai J, Sun X, Geracioti TD, Hamner MB, Lohr J, Rosse R, Summerall L, Naylor JC, Cusin C, Lang AJ, Raman R, Stein MB. A randomized controlled trial of ganaxolone in posttraumatic stress disorder. Psychopharmacology (Berl). 2017 Aug;234(15):2245-2257. doi: 10.1007/s00213-017-4649-y. Epub 2017 Jul 1. PMID 28667510

RESULTS

PARTICIPANT FLOW:
Groups:
- Ganaxolone: active
  Ganaxolone: 200-600 milligram (mg) twice daily (bid), capsules, up to 12 weeks
Period: Overall Study
Arm/Group | Ganaxolone | Placebo
Started | 59 | 53
Completed | 42 | 44
Not Completed | 17 | 9
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 9 | 3
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Noncompliance | 1 | 0
Not completed — Relocated out of area | 0 | 1
Not completed — Other | 2 | 2
Not completed — multiple reasons | 1 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-treat (mITT) Population: Included randomized participants who had been dispensed study medication and had at least one post-Baseline data point during the 6-week placebo-controlled blinded phase of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ganaxolone | Placebo | Total
Number analyzed (Participants) | 59 | 53 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.78 (10.54) | 37.74 (10.86) | 38.29 (10.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 24
  Male | 44 | 44 | 88
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 50 | 48 | 98
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 16 | 35
  White | 30 | 35 | 65
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Clinician-Administered Posttrautamtic Stress Disorder (PTSD) Scale (CAPS) to Week 6
Description: The CAPS was a structured interview that queries participants about each of the 17 Diagnostic and Statistical manual of Mental Disorders IV (DSM-IV) criteria B, C, and D symptoms of PTSD. Each item has a frequency score (0-4) and intensity score (0-4). The CAPS total score is the sum of frequency and intensity ratings for each item and the score range was 0: no symptoms to 136: severe symptoms. Higher score indicates worse symptoms. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Week 0) and at Week 2, Week 4 and Week 6
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Placebo: non-active Placebo: capsules, bid, up to 12 weeks
- Ganaxolone: active Ganaxolone: 200-600 mg bid, capsules, up to 12 weeks
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 50 | 49
Scores on a scale
  Week 2 | 65.78 (24.4) | 62.67 (21.39)
  Week 4: number analyzed (Participants) | 46 | 43
  Week 4 | 63.2 (23.06) | 61.30 (23.42)
  Week 6: number analyzed (Participants) | 44 | 42
  Week 6 | 60.64 (27.54) | 54.05 (25.86)

2. Secondary Outcome: Change From Baseline in PTSD Re-Experience Score
Description: The CAPS was a structured interview that queries participants about each of the 17 Diagnostic and Statistical manual of Mental Disorders IV (DSM-IV) criteria B, C, and D symptoms of PTSD. Each item has a frequency score (0-4) and intensity score (0-4). The Re-experience score is the sum of frequency and intensity ratings for items from cluster B and the score range was 0: no symptoms to 40: severe symptoms. Higher score indicates worse symptoms. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Week 0) and at Week 2, Week 4 and Week 6
Population: mITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 50 | 49
Scores on a scale
  Week 2 | 16.56 (10.61) | 14.45 (8.98)
  Week 4: number analyzed (Participants) | 46 | 43
  Week 4 | 16.54 (8.03) | 14.16 (8.83)
  Week 6: number analyzed (Participants) | 44 | 42
  Week 6 | 15.5 (11.11) | 12.31 (9.28)

3. Secondary Outcome: Change From Baseline in PTSD Avoidance Score
Description: The CAPS was a structured interview that queries participants about each of the 17 Diagnostic and Statistical manual of Mental Disorders IV (DSM-IV) criteria B, C, and D symptoms of PTSD. Each item has a frequency score (0-4) and intensity score (0-4). The Avoidance score is the sum of frequency and intensity ratings for items from cluster C.and the score range was 0: no symptoms to 56: severe symptoms. Higher score indicates worse symptoms. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Week 0) and at Week 2, Week 4 and Week 6
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 50 | 49
Scores on a scale
  Week 2 | 27.06 (11.54) | 26.29 (10.76)
  Week 4: number analyzed (Participants) | 46 | 43
  Week 4 | 25.87 (11.69) | 26.09 (11.87)
  Week 6: number analyzed (Participants) | 44 | 42
  Week 6 | 24.82 (11.45) | 23.52 (13.1)

4. Secondary Outcome: Change From Baseline in PTSD Hyperarousal Score
Description: The CAPS was a structured interview that queries participants about each of the 17 Diagnostic and Statistical manual of Mental Disorders IV (DSM-IV) criteria B, C, and D symptoms of PTSD. Each item has a frequency score (0-4) and intensity score (0-4). The Hyperarousal score is the sum of frequency and intensity ratings for items from cluster D and the score range was 0: no symptoms to 40: severe symptoms. Higher score indicates worse symptoms. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Week 0) and at Week 2, Week 4 and Week 6
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 50 | 49
Scores on a scale
  Week 2 | 22.16 (7.73) | 21.94 (7.76)
  Week 4: number analyzed (Participants) | 46 | 43
  Week 4 | 20.78 (7.8) | 21.05 (8.48)
  Week 6: number analyzed (Participants) | 44 | 42
  Week 6 | 20.32 (9.07) | 18.21 (8.55)

5. Secondary Outcome: Number of Participants With Response to Clinical Global Impression - Improvement (Investigator) (CGI-II) Scale
Description: The CGI-II scale is a 7-point scale where the investigator was required to assess how much the participant's illness has improved or worsened relative to a Baseline state at the beginning of the intervention, and rated as 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. Higher score indicated worse symptoms. The score was grouped into two categories for analysis: Responders=1 or 2, Non-responders=3-7.
Time Frame: Week 2, Week 4 and Week 6
Population: mITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 49 | 48
Participants
  Week 2 - Non-Responder | 42 | 45
  Week 2 - Responder | 7 | 3
  Week 4 - Non-Responder: number analyzed (Participants) | 46 | 43
  Week 4 - Non-Responder | 37 | 38
  Week 4 - Responder: number analyzed (Participants) | 46 | 43
  Week 4 - Responder | 9 | 5
  Week 6 - Non-Responder: number analyzed (Participants) | 44 | 41
  Week 6 - Non-Responder | 32 | 27
  Week 6 - Responder: number analyzed (Participants) | 44 | 41
  Week 6 - Responder | 12 | 14

6. Secondary Outcome: Number of Participants With Response to CGI-I Subject Scale Clinical Global Impression - Improvement (Subject) (CGI-IS) Scale
Description: The CGI-IS scale is a 7-point scale where the participant assesses how much the illness has improved or worsened relative to a Baseline state at the beginning of the intervention, and rated as 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. Higher score indicated worse symptoms. The score was grouped into two categories for analysis: Responders=1 or 2, Non-responders=3-7.
Time Frame: Week 2, Week 4 and Week 6
Population: mITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 50 | 48
Participants
  Week 2 - Non-Responder | 45 | 46
  Week 2 - Responder | 5 | 2
  Week 4 - Non-Responder: number analyzed (Participants) | 46 | 43
  Week 4 - Non-Responder | 39 | 37
  Week 4 - Responder: number analyzed (Participants) | 46 | 43
  Week 4 - Responder | 7 | 6
  Week 6 - Non-Responder: number analyzed (Participants) | 44 | 42
  Week 6 - Non-Responder | 37 | 37
  Week 6 - Responder: number analyzed (Participants) | 44 | 42
  Week 6 - Responder | 7 | 5

7. Secondary Outcome: Change From Baseline in PTSD Checklist (PCL) Scores
Description: The PCL is a 17-item self-report scale representing all DSM-IV criteria for PTSD, including re-experiencing, avoidance and numbing, and hyperarousal criteria. Each item is scored 1-5 (1=not at all; 2=a little bit; 3=moderately; 4=quite a bit; 5=extremely). The total score is the sum of 17 item scores and ranged from 17: no symptoms to 85: severe symptoms. Higher score indicated worse symptoms. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Week 0) and at Week 2, Week 4 and Week 6
Population: mITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 50 | 49
Scores on a scale
  Week 2 | 54.4 (14.24) | 50.79 (15.05)
  Week 4: number analyzed (Participants) | 46 | 43
  Week 4 | 52.93 (15.31) | 48.74 (16.2)
  Week 6: number analyzed (Participants) | 44 | 42
  Week 6 | 51.75 (15.73) | 46.33 (17.29)

8. Secondary Outcome: Change From Baseline in Profile of Mood States (POMS) Total Score
Description: The POMS is a factor-analytically derived 65 item self-report inventory with 5-point measures of five dimensions of negative mood: anger/irritability, anxiety/tension, depression/dejection, confusion/bewilderment, and fatigue/inertia, as well as vigor/activity. Total score was calculated as Fatigue + Mood (sum [Confusion, anger, Anxiety/Tension, Depression])- Vigor. Score ranged from 0: no symptoms to 200: severe symptoms; higher score indicated worse symptoms. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Week 0) and Week 6
Population: mITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 45 | 42
Scores on a scale | 80.07 (50.21) | 66.98 (45.29)

9. Secondary Outcome: Change From Baseline in Patient Health Questionnaire (PHQ-9) Score
Description: The PHQ-9 is the nine-item depression scale of the Patient Health Questionnaire. The nine items of the PHQ-9 are based directly on the nine diagnostic criteria for major depressive disorder in the DSM-IV. Each item is scored 0-3 (0=not at all; 1=several days; 2=more than half the days; 3= nearly every day). The total score is the sum of 9 item scores and ranged 0: no depression to 27: severe depression. The higher the total score, the worse the depression. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Week 0) and Week 6
Population: mITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 46 | 45
Scores on a scale | 12.13 (7.47) | 10.71 (6.99)

10. Secondary Outcome: Change From Baseline in Insomnia Severity Index (ISI) Score
Description: The ISI is a self-rated questionnaire assessing the difficulty over the past two weeks with falling to sleep, awakening in the middle of the night, and early morning awakening, as well as the degree to which insomnia impairs daily function. It included 5 items (rst item has 3 sub-questions), so a total of 7 questions. Each question is scored 0-4 (0=none, 1=mild, 2=moderate, 3=severe, 4=very severe). The total score is the sum of 7 item scores and ranged from 0: no symptoms to 28: severe symptoms. Higher score indicated worse symptoms. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline (Week 0) and Week 6
Population: mITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 46 | 45
Scores on a scale | 17.04 (7.69) | 14.36 (7.94)

11. Secondary Outcome: Change From Baseline in Connor-Davidson Resilience Scale (CD-RISC) Score
Description: The CD-RISC comprises 25 items, each rated on a 5-point scale (0-4), with higher scores reflecting greater resilience that may be a target for treatment in stress disorders. The total score is the sum of 25 item scores and ranged from 0: no symptoms to 100: worse symptoms. Higher score indicates worse symptoms. Baseline was defined as the Day 0 assessment before study drug infusion. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value
Time Frame: Baseline (Week 0) and Week 6
Population: mITT Population. Only those participants with data available at the specified data points were analyzed
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | Ganaxolone
Number analyzed (Participants) | 45 | 44
Scores on a scale | 60.84 (20.67) | 61.01 (19.56)

ADVERSE EVENTS:
Time Frame: Up to Week 15
Arm/Group | Ganaxolone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/53
Serious Adverse Events (participants affected / at risk) | 3/59 | 0/53
Other Adverse Events (participants affected / at risk) | 39/59 | 32/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=59) | Placebo (N=53)
Suicidal Ideation (Psychiatric disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Confusion (Nervous system disorders) | 1 | 0
Balance Issues (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ganaxolone (N=59) | Placebo (N=53)
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Dry Eye (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 4 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 1 | 1
Fatigue (Gastrointestinal disorders) | 5 | 2
Feeling drunk (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Irritability (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Sensation of pressure (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Inadequate analgesia (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 0 | 1
Blood urine present (Investigations) | 1 | 1
Liver function test abnormal (Investigations) | 1 | 0
Protein urine present (Investigations) | 1 | 0
Tandem galt test abnormal (Investigations) | 1 | 0
Weight increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Ataxia (Nervous system disorders) | 2 | 0
Balance disorder (Nervous system disorders) | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 4 | 0
Dysarthria (Nervous system disorders) | 3 | 0
Headache (Nervous system disorders) | 8 | 4
Lethargy (Nervous system disorders) | 2 | 1
Migraine (Nervous system disorders) | 1 | 0
Motor dysfunction (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Sedation (Nervous system disorders) | 5 | 4
Slow speech (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 11 | 7
Tremor (Nervous system disorders) | 2 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0
Anger (Psychiatric disorders) | 1 | 0
Anorgasmia (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 0
Depressed mood (Psychiatric disorders) | 0 | 1
Depressed (Psychiatric disorders) | 1 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0
Initial insomnia (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 2
Nightmare (Psychiatric disorders) | 4 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 2
Psychomotor retardation (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1
Tic (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Upper airway resistance syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Suicide of companion (Social circumstances) | 1 | 0
Product used for unknown indication (Surgical and medical procedures) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No